CLINICAL TRIAL: NCT01446627
Title: Comparison of Vicryl Absorbable Sutures and Metal Staples Used in Skin Closure Following Cesarean Section
Brief Title: Use of Insorb Absorbable Vicryl Staples in Skin Closure for Cesarean Section
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jonathan P Faro, Assistant Professor, ObGyn, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-GEN-11-0169
Record Dates: First submitted 2011-09-30; First posted 2011-10-05 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Wound Infection
Keywords: Absorbable vicryl subcuticular staples; metal staples; wound healing; cesarean section
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- metal staples
  Interventions: Other: There is no intervention for this study
- Insorb vicryl staples
  Interventions: Other: There is no intervention for this study

INTERVENTIONS:
Other: There is no intervention for this study — None, no intervention made.
  Other Names: This is an observational study, involving human subjects. It is a clinical study, but not a clinical trial. No intervention will be made.

SUMMARY:
The purpose of this study is to evaluate the incidence of wound breakdown or wound infection following skin closure with Insorb subcuticular absorbable staples versus metal staples after cesarean section through a retrospective chart analysis.

DETAILED DESCRIPTION:
Procedures:

A list will be compiled of patients who underwent cesarean section at Memorial Hermann Hospital in the Texas Medical Center from January 1st 2010 through January 1st 2011. Only UT patients who had their skin closed with Insorb or metal staples will be included in this list. Patients' clinical charts will be reviewed for post-operative follow-up, and notes will be made of the wound assessment. Any complications such as infection, seroma, hematoma, and wound separation or delayed healing will be recorded. Additional notes will be made of any co-morbid conditions, including, but not limited to, >30 BMI, chronic hypertension, diabetes mellitus, HIV, history of tobacco use.

Once the data is gathered, it will be compared with published national averages to determine if there is an increased risk of wound separation or wound infection at our institution. In addition, rated of infection and wound breakdown following closure with either absorbable or metal staples will be compared by Fisher's exact test, to determine statistical significance.

Course of Study: Data will be obtained from UT patients who underwent cesarean section from January 1st, 2010 through January 1st, 2011. Only patients who had skin closure with InSorb or metal staples will be included in analysis.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean sections
* UT patients

Exclusion Criteria:

* Patients who have skin closed with suture, per attending choice.

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women undergoing cesarean section who have their skin incision closed with staples.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Wound infection/separation | from time of surgery up until wound assessed to be completely healed, no longer than 1 year.

SECONDARY OUTCOMES:
wound hematoma | From time of surgery up until wound assessed to be completely healed, no longer than 1 year.
wound seroma | From time of surgery up until wound assessed to be completely healed, no longer than 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Faro, MD, PhD, Principal Investigator — UTHSC at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States